CLINICAL TRIAL: NCT04159948
Title: Preoperative Carbohydrate Drink Prior to Elective Caesarean Section: A Randomized Controlled Trial.
Brief Title: Preoperative Carbohydrate Drink Prior to Elective Caesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Coombe Women and Infants University Hospital (Other)
Responsible Party: Principal Investigator, Ruairi Irwin, Anaesthesia SpR, Coombe Women and Infants University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CWIUH-CHO (16-2019)
Record Dates: First submitted 2019-11-08; First posted 2019-11-12 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Fasting; Cesarean Delivery Affecting Fetus; Glucose, Low Blood
Keywords: Carbodydrate drink
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Intervention Model Description: 3 arms with equal allocation.
Who Masked: Outcomes Assessor
Masking Description: Patient will not be blinded to which arm they have been allocated to. Outcome assessors will be unaware of group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Water (Placebo Comparator): Patients will be allowed to drink water up to 2 hours before their caesarean section.
  Interventions: Dietary Supplement: Carbohydrate drink
- Carbohydrate drink (Active Comparator): Patients will be allowed to drink a designated carbohydrate drink up to 2 hours before their caesarean section.
  Interventions: Dietary Supplement: Carbohydrate drink
- Apple juice (Active Comparator): Patients will be allowed to drink apple juice up to 2 hours before their caesarean section.
  Interventions: Dietary Supplement: Carbohydrate drink

INTERVENTIONS:
Dietary Supplement: Carbohydrate drink — This is a commercially available "pre-op" carbohydrate drink used in enhanced recovery programmes.

SUMMARY:
Prior to caesarean section, patients should fast from solid food for 6 hours and from clear fluids for 2 hours. Carbohydrate drinks can also be consumed up to 2 hours before surgery. These drinks have been shown to improve patient well-being after surgery and may potentially improve the neonatal blood glucose level after delivery and reduce the risk of a low blood glucose level. This study aims to assess the influence of pre-operative carbohydrate drinks on blood glucose levels of the baby at delivery.

DETAILED DESCRIPTION:
Patients recruited to the study will be randomised to one of 3 groups.

Group 1 will receive standard care as per our current practice. This includes fasting from solids for 6 hours prior to surgery and clear fluids for up to 2 hours prior to surgery.

Group 2 will receive a carbohydrate (CHO) drink preoperatively as well as adhering to standard care. Patients will be allowed to drink this CHO drink as required from admission to hospital on the morning of their surgery. They will also receive a further 400ml bolus at 2 hours prior to surgery.

Group 3 will receive an apple juice drink preoperatively as well as adhering to standard care. Patients will be allowed to drink this apple juice drink as required from admission to hospital on the morning of their surgery. They will also receive a further 400ml bolus at 2 hours prior to surgery.

Before the start of surgery, the patients non-dominant hand grip strength will be assessed using the dynamometer. Their subjective sense of thirst and hunger will be assessed. Their fasting times for food and fluids will be recorded. The patients' blood glucose will be measured from a blood sample as their intravenous cannula is inserted. The maternal urinary ketones will be measured from a urine sample upon insertion.

The neonatal blood cord glucose will be measured from both an arterial and venous cord blood sample after delivery. This will be performed by the trained anaesthesia research fellow. Should hypoglycemia be identified, the hospital's neonatal hypoglycemia algorithm will be followed appropriately.

The patients will be followed up at 24 hours by an outcome assessor blinded to the group allocation. Numerical rating scale (NRS) pain scores, postoperative nausea and vomiting and quality of recovery will be assessed at the patients beside. All neonates will be followed up to calculate admissions to neonatal unit and the number of glucose sachets required for hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Elective caesarean section for singleton pregnancy under neuraxial anaesthesia.
* Subjects able to give informed consent and willing to comply with the study protocol.
* Subjects must be greater than 18 years old.

Exclusion Criteria:

* Diabetes Mellitus - including gestational diabetes.
* Known foetal abnormality.
* General anaesthesia.
* Gestation < 37 weeks.
* Steroids received within 4 days of delivery.
* Low birth weight 2.5 kg (IUGR)
* BMI > 40 kg/m2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-08-10 (Estimated); Study Completion 2021-08-10 (Estimated)

PRIMARY OUTCOMES:
Neonatal cord blood glucose | 0 hours
  A blood sample of the neonatal cord will be checked immediately after delivery.

SECONDARY OUTCOMES:
Neonate tolerating 1st oral feeding. | 0-2 hours
  Binary outcome - Neonate consuming adequate breast or bottle milk.
Number of neonatal rescue oral glucose sachets given. | 6 hours
  Continuous - Number of neonatal rescue oral glucose sachets given.
Neonate requiring ICU admission and treatment for hypoglycemia | 6 hours
  Binary - Neonate requiring ICU admission and treatment for hypoglycemia
Maternal blood glucose | 0 hours
  Maternal blood glucose prior to the start of caesarean section.
Maternal urinary ketones | 0 hours
  Maternal urinary ketones prior to the start of caesarean section.
Maternal subjective sense of thirst prior to the start of caesarean section. | 0 hours
  Scored on a scale 0-10
Maternal subjective sense of hunger prior to the start of caesarean section. | 0 hours
  Scored on a scale 0-10
Maternal quality of recovery | 24 hours
  Measured using the ObsQoR-11 questionnaire
Resumption of oral diet post caesarean section. | 24 hours
  Time until resumption of oral diet
Resumption of fluids post caesarean section. | 24 hours
  Time until resumption of fluids
Post-operative nausea and vomiting (PONV) | 24 hours
  The self reported incidence of PONV
PONV requiring treatment | 24 hours
  PONV requiring pharmacological treatment
Pain scores | 24 hours
  Pain scores at rest and movement on scale 0-10
Breastfeeding success | 24 hours
  Binary - whether continuing attempted breast feeding at 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Terry Tan, Study Director — Head of Department of Anaesthesia CWIUH
Locations (1):
- Coombe Women and Infants University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided